CLINICAL TRIAL: NCT02888262
Title: The Bipolar Illness Onset Study (the BIO Study)
Acronym: BIO
Status: Active, not recruiting | Type: Observational
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Lars Vedel Kessing, Professor, MD, DMSc., Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Other Study IDs: Psychiatric Center Copenhagen
Record Dates: First submitted 2016-08-24; First posted 2016-09-02 (Estimated); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Bipolar Disorder
Keywords: Bipolar disorder; Blood; Smartphone; Brain imaging; Cognition; Neuropsychology
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Urine Hair
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients with bipolar disorder: Patients with newly diagnosed bipolar disorder
- Healthy first generation relatives: Healthy first generation relatives to the included patients
- Healthy individuals: Healthy individuals without a family history of psychiatric disorders

SUMMARY:
This longitudinal study aims to identify 1) a composite blood-based biomarker, 2) a composite electronic Smartphone-based biomarker and 3) a neurocognitive signature for bipolar disorder

DETAILED DESCRIPTION:
The study will include 300 patients with newly diagnosed/first episode bipolar disorder, 200 healthy siblings or child family members and 100 healthy individuals without a family history of affective disorder. All individuals will be investigated with repeated blood tests, Smartphone recordings, neuropsychological tests and brain imaging during a five to ten year study period.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed/first episode bipolar patients,
2. First-generation relatives (siblings and children aged 15 to 40 years) to the recruited newly diagnosed/first episode bipolar patients.
3. Age- and gender matched sample of healthy individuals without a first-generation family history of effective disorders

Exclusion Criteria:

1. Significant physical disorders
2. Schizophrenia or related disorders

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. 300 patients referred to the Copenhagen Affective Disorder Clinic as newly diagnosed/first episode bipolar patients, i.e., onset of first manic or hypomanic episode or when the diagnosis of bipolar disorder is made for the first time.
  2. 200 first-generation relatives (siblings and children aged 15 to 40 years) to the recruited newly diagnosed/first episode bipolar patients.
  3. 100 age-, gender- and IQ-matched sample of healthy individuals without a first-generation family history of affective disorders recruited among blood donors from the Blood Bank at Rigshospitalet, Copenhagen, as in prior studies.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Composite blood based biomarker | 5 years

SECONDARY OUTCOMES:
Composite smartphone based biomarker including self reported and smartphone generated data | 5 years
  Composite smartphone based biomarker including 1) self reported data and 2) smartphone generated data on physical activity 3) social activity and 4) voice features collected during phone calls
Composite neurocognitive marker including "Cold" and "Hot" cognition. | 5 years
  Composite neurocognitive marker including "Cold" cognition assessed with neuropsychological tests probing verbal memory and executive function and "Hot" cognition assessed with a comprehensive computerized battery of cognitive tests probing (i) emotional processing (ii) reward processing and (iii) emotional regulation.

CONTACTS AND LOCATIONS:
Overall Officials: Lars V Kessing, Professor, Principal Investigator — Psychiatric Center Copenhagen
Locations (1):
- Psychiatric Center Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stanislaus S, Coello K, Kjaerstad HL, Sletved KSO, Seeberg I, Frost M, Bardram JE, Jensen RN, Vinberg M, Faurholt-Jepsen M, Kessing LV. Prevalences of comorbid anxiety disorder and daily smartphone-based self-reported anxiety in patients with newly diagnosed bipolar disorder. Evid Based Ment Health. 2021 Nov;24(4):137-144. doi: 10.1136/ebmental-2021-300259. Epub 2021 Jun 3. PMID 34083204
- [Derived] Stanislaus S, Vinberg M, Melbye S, Frost M, Busk J, Bardram JE, Kessing LV, Faurholt-Jepsen M. Smartphone-based activity measurements in patients with newly diagnosed bipolar disorder, unaffected relatives and control individuals. Int J Bipolar Disord. 2020 Nov 2;8(1):32. doi: 10.1186/s40345-020-00195-0. PMID 33135120
- [Derived] Stanislaus S, Vinberg M, Melbye S, Frost M, Busk J, Bardram JE, Faurholt-Jepsen M, Kessing LV. Daily self-reported and automatically generated smartphone-based sleep measurements in patients with newly diagnosed bipolar disorder, unaffected first-degree relatives and healthy control individuals. Evid Based Ment Health. 2020 Nov;23(4):146-153. doi: 10.1136/ebmental-2020-300148. Epub 2020 Aug 24. PMID 32839276
- [Derived] Melbye SA, Stanislaus S, Vinberg M, Frost M, Bardram JE, Sletved K, Coello K, Kjaerstad HL, Christensen EM, Faurholt-Jepsen M, Kessing LV. Mood, activity, and sleep measured via daily smartphone-based self-monitoring in young patients with newly diagnosed bipolar disorder, their unaffected relatives and healthy control individuals. Eur Child Adolesc Psychiatry. 2021 Aug;30(8):1209-1221. doi: 10.1007/s00787-020-01611-7. Epub 2020 Aug 2. PMID 32743692
- [Derived] Kessing LV, Munkholm K, Faurholt-Jepsen M, Miskowiak KW, Nielsen LB, Frikke-Schmidt R, Ekstrom C, Winther O, Pedersen BK, Poulsen HE, McIntyre RS, Kapczinski F, Gattaz WF, Bardram J, Frost M, Mayora O, Knudsen GM, Phillips M, Vinberg M. The Bipolar Illness Onset study: research protocol for the BIO cohort study. BMJ Open. 2017 Jun 23;7(6):e015462. doi: 10.1136/bmjopen-2016-015462. PMID 28645967